CLINICAL TRIAL: NCT02065661
Title: Product Validation Study of 2 New Devices, EZ-NG (RightSpot pH Indicator) and EZ-pH (RightLevel pH Indicator)
Status: Completed | Type: Observational
Sponsor: Florida Hospital Tampa Bay Division (Other)
Responsible Party: Sponsor
Other Study IDs: EZ Product Validation Study
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Small Bowel Obstruction; Colectomy; Bowel Surgeries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EZ Holdco Inc. has developed two devices for the measurement of gastric content pH. The devices, EZ-NG and EZ-pH, rapidly check gastric pH by aspirating gastric contents into the device through a nasogastric (NG) tube and causing a color change in the device. The color change is then compared to the reference indicator on the device to determine a pH value of the aspirate. Currently there is no bedside rapid way to check gastric pH that protects the clinician from being exposed to the aspirate.

1. Primary Objective To assess the accuracy of the pH measurement of gastric fluid on the devices by comparing the reading on the 2 devices to a standard clinically approved pH probe.
2. Secondary Objective To determine what percentage of time the EZ-NG - RightSpot pH indicator could have been used to determine proper placement of the NG tube when initially placed.

ELIGIBILITY:
Inclusion Criteria:

* Consented elective surgical patient

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consented elective surgical candidates
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
1. Primary Objective To assess the accuracy of the pH measurement of gastric fluid on the devices by comparing the reading on the 2 devices to a standard clinically approved pH probe. | 60 min

SECONDARY OUTCOMES:
2. Secondary Objective To determine what percentage of time the EZ-NG - RightSpot pH indicator could have been used to determine proper placement of the NG tube when initially placed. | 60 min